CLINICAL TRIAL: NCT07199868
Title: PRP Group & Control Group in Poseidon Poor Responders
Brief Title: The Role of Ovarian PRP Therapy in Poseidon Poor Responders Women Undergoing ICSI Cycle
Acronym: PRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karbala University (Other)
Responsible Party: Principal Investigator, Itlal Asadi, Principal Investigator, Karbala University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0009-0007-1354-0259; non (Other: non)
Record Dates: First submitted 2025-09-09; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Poor Ovarian Reserve; Platelet Derived Growth Factor
MeSH Terms: interventions — Conscious Sedation

STUDY DESIGN:
Intervention Model Description: During early-mid follicular phase, using TV-US guidance and conscious sedation, 1.5 ml of PRP was injected into each ovary's subcortical layer using a 17-gauge ovum pick-up needle.
Masking Description: non
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ovarian PRP injection in poor responders (Experimental): During early-mid follicular phase, using TV-US guidance and conscious sedation, 1.5 ml of PRP was injected into each ovary's subcortical layer using a 17-gauge ovum pick-up needle.
  Interventions: Procedure: During early-mid follicular phase, using TV-US guidance and conscious sedation, 1.5 ml of PRP was injected into each ovary's subcortical layer using a 17-gauge ovum pick-up needle.

INTERVENTIONS:
Procedure: During early-mid follicular phase, using TV-US guidance and conscious sedation, 1.5 ml of PRP was injected into each ovary's subcortical layer using a 17-gauge ovum pick-up needle. — During early-mid follicular phase, using TV-US guidance and conscious sedation, 1.5 ml of PRP was injected into each ovary's subcortical layer using a 17-gauge ovum pick-up needle.

SUMMARY:
Objective : This study aims to evaluate the impact of ovarian PRP therapy compared to control in Poseidon females undergoing ICSI cycles.

Material and Methods: A randomized controlled trial was conducted from Jan 2024 to Feb 2025, involving 102 Poseidon women, Participants were divided into a PRP group (n=50), who received ovarian PRP injections and a control group (n=52), who received no PRP. All participants underwent ICSI cycles, embryological and pregnancy outcomes were compared between both groups within each Poseidon group.

DETAILED DESCRIPTION:
2. Materials And Methods 2.1. Study design This study was conducted at a private fertility center in Karbala, Iraq, from Jan 2024 to Feb 2025. All participants provided written informed consent prior to enrollment, and ethical approval was obtained from the College of Medicine, Karbala University (reference number 25-8).

2.2. Participants A total of 102 Poseidon POR women were enrolled where Inclusion criteria were infertile Poseidon groups 2, 3, 4 women with no history of chronic illness or pelvic pathology. All male partners were either normozoospermic or had mild OAT delivered fresh ejaculated samples for ICSI.

Exclusion criteria were ovarian failure due to sex chromosome abnormalities, current use of anticoagulants and history of bleeding disorders. Participants were assigned into two groups: Study group (n=50), who underwent ovarian PRP injections once or twice times within six months prior to ICSI cycle, and control group (n=52), who did not receive PRP therapy.

2.3. PRP preparation and injection Twenty mL of peripheral blood was drawing under sterile conditions using Lora PRP tubes (Modern Technology Company). Frist the blood was centrifuged at 1600 rpm for 10 minutes (soft spin). Then the plasma and superficial buffy coat were transferred into a sterile tube containing no anticoagulant and centrifuged again at 3500 rpm for 5 minutes (hard spin). The upper 2/3rd (platelet-poor plasma, PPP) were discarded, and the platelet pellets were homogenized in the lower 1/3rd of plasma to create 3 mL of platelets concentrate of 3-5 times higher than basal and injected within one hour of preparation (11). During early-mid follicular phase, using TV-US guidance and conscious sedation, 1.5 ml of PRP was injected into each ovary's subcortical layer using a 17-gauge ovum pick-up needle. A second PRP injection was administered when subsequent ORTs (AMH,AFC) and hormone levels (FSH, LH, E2) showed suboptimal results in patient's next menstrual cycles.

2.4. ICSI cycle outcomes All patients starting same COS protocol began on CD3 using (300-450 iu) of Gonal-F (r-FSH); Merck ± (u-HMG);LG in flexible antagonist protocol, (Cetrotide); Merck. Final oocyte maturation was triggered by 250 mcg r-hCG (Ovitrelle; Serono) ± 0.2 mg GnRH agonist (Decapeptyl; Merck) 35 hours before oocyte retrieval when dominant follicles reached (17-18) mm. Embryological outcomes including; MII oocytes, embryos quantity and quality were compared in both group. In all embryo transfer cycles, 2-4 embryos grade A± B of age 2-5 day were transferred. The clinical outcomes included pregnancy rate (serum β-HCG ≥100 mIU/mL), miscarriage rate (the loss of a pregnancy before 24 weeks), Live Birth rates (delivery of a living baby after 24 weeks) and overall cycle outcomes were compared in both groups.

ELIGIBILITY:
Inclusion Criteria:

1 - infertile Poseidon groups 2, 3, 4 women 2- no history of chronic illness or pelvic pathology. 3- All male partners were either normozoospermic or had mild OAT delivered fresh ejaculated samples for ICSI.

Exclusion Criteria:

1 - ovarian failure due to sex chromosome abnormalities, 2- current use of anticoagulants 3- history of bleeding disorders.

Ages: 21 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 102 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
numbers of Meta phase II oocytes and embryos post ovarian PRP | one year
  Primary embryological outcomes including; metaphase II oocytes and embryos numbers in addition to their quality post ovarian PRP were compared in both study & control groups

CONTACTS AND LOCATIONS:
Overall Officials: Itlal J AL Asadi, MD, Principal Investigator — Department of Obstetrics & Gynecology, College of Medicine, Karbala University
Locations (2):
- Iraq (2):
  - Collage of medicine, Baghdad
  - Collage of medicine, Karbala

IPD SHARING:
Plan to Share IPD: Undecided
on request only

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: The role of Ovarian PRP Therapy (2025-01-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT07199868/Prot_SAP_000.pdf
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: ICSI Cycles (2025-01-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT07199868/Prot_SAP_ICF_001.pdf
  • Informed Consent Form: Poseidon Poor Responders (2025-01-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT07199868/ICF_002.pdf